CLINICAL TRIAL: NCT02542241
Title: Hypertonic Saline Resuscitation for Early Closure of Open Abdomen in Trauma Patients
Brief Title: Hypertonic Saline Resuscitation in Trauma Patients After Hemorrhage Control
Acronym: CELTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funds to continue recruitment
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Alberto Federico García, MD., Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00877
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Abdominal Injuries
Keywords: Open abdomen; hypertonic saline solution; intensive care
MeSH Terms: conditions — Abdominal Injuries | interventions — Sodium Chloride; Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Chloride [3%] (Experimental)
  Interventions: Drug: Sodium Chloride [3%]
- Sodium Chloride [0.9%] (Active Comparator)
  Interventions: Drug: Sodium Chloride [0.9%]

INTERVENTIONS:
Drug: Sodium Chloride [3%] — Patients in this arm will receive an intravenous infusion of 3% hypertonic saline at a 50 cc/hour rate, which will be administered by an infusion pump during the first 72 hours after the damage control surgery. A total of 3600cc will be administered throughout 72 hours ( 1200cc every 24 hours).
  Other Names: Hypertonic Saline Solution; NaCl
  Arms: Sodium Chloride [3%]
Drug: Sodium Chloride [0.9%] — Patients in this arm will receive an intravenous infusion of 0.9% hypertonic saline at a 50 cc/hour rate, which will be administered by an infusion pump during the first 72 hours after the damage control surgery. A total of 3600cc will be administered throughout 72 hours ( 1200cc every 24 hours).
  Other Names: Physiologic Saline Solution; Normal Saline
  Arms: Sodium Chloride [0.9%]

SUMMARY:
This study aimed to determine whether hypertonic saline solution is effective in the resuscitation of injured patients undergoing abdominal damage control surgery regarding early closure of the abdominal wall.

DETAILED DESCRIPTION:
A double-blind, controlled, randomized clinical trial was conducted to determine the impact of an infusion of hypertonic saline 3% vs. isotonic saline 0.9% at a dose of 50 mL/hr for the first 72 hours in patients with abdominal trauma requiring damage control surgery regarding some clinically relevant outcomes. These outcomes were: The timing of abdominal cavity closure, fluids balance, abdominal hypertension, and abdominal compartment syndrome occurrence, organ dysfunction, and 28 days' mortality.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal trauma requiring damage control surgery.
* Acceptance by the patient or by a proxy to be included in the trial.

Exclusion Criteria:

* Concomitant severe head trauma, defined by a Glasgow score <9, before receiving sedation or by the presence of cerebral edema or intracranial injury on a CT-scan.
* Pregnancy
* Patient not included 4 hours or more after damage control surgery.
* Damage control laparotomy performed for other indications other than trauma.
* Not index damage control laparotomy
* No acceptance to participate in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-11-27; Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Abdominal wall closure | 7 days
  Proportion of patients in which closure of abdominal wall was achieved in the first 7 days after injury.

SECONDARY OUTCOMES:
Fluid Balance measured in cm3 | 72 hours
  Fluid balance during the first 72 hours after injury.
  Defined as the difference between the amount of fluids taken into the body and the amount excreted or lost. Input includes oral fluids, infused intravenous fluids and blood products. Output includes fluid loss as urine, emesis and wound drainage among others.
Incidence of Abdominal compartment syndrome | 7 days
  Incidence of abdominal compartment syndrome (defined as sustained intra-abdominal pressure > 20 mmHg, accompanied by new organ dysfunction, defined as a score > 2, under the SOFA scale compromising lung, kidney, or heart) during the first 7 days after injury.
Incidence of Organ Failure | 7 days
  Incidence of organ failure (defined as SOFA score greater than 2).
Mortality | 28 days
  28 day mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Alberto F García, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Clinica Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
The individual participant data contained in the datasets generated and/or analyzed for the current study are not publicly available as recommended by the local ethical and research committee involving human beings (Fundación Valle del Lili, Cali, Colombia) but could be available from the corresponding author on reasonable request and under prior approval by such committee.

REFERENCES:
- [Derived] Garcia AF, Manzano-Nunez R, Carrillo DC, Chica-Yanten J, Naranjo MP, Sanchez AI, Mejia JH, Ospina-Tascon GA, Ordonez CA, Bayona JG, Puyana JC. Hypertonic saline infusion does not improve the chance of primary fascial closure after damage control laparotomy: a randomized controlled trial. World J Emerg Surg. 2023 Jan 9;18(1):4. doi: 10.1186/s13017-023-00475-x. PMID 36624448